CLINICAL TRIAL: NCT04168541
Title: Plasma Glucose and Insulin Response to Six Oral Nutrition Supplements in Persons With Type 2 Diabetes Mellitus
Brief Title: Glycemic Response in Persons With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17.11.US.HCN
Record Dates: First submitted 2018-02-01; First posted 2019-11-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This will be a randomized crossover design. The subjects will be randomized to one of six interventions on six separate study days, one week apart.
Who Masked: Participant
Masking Description: Study staff will not be blinded to product assignment. Study participants will be blinded to product assignment. Product will be provided in unlabeled plastic cups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Oral Nutrition Supplement A (Active Comparator): Product containing calories from carbohydrate, protein, and fat
  Interventions: Other: Oral Nutrition Supplement
- Oral Nutrition Supplement B (Active Comparator): Product containing calories from carbohydrate, protein, and fat
  Interventions: Other: Oral Nutrition Supplement
- Oral Nutrition Supplement C (Active Comparator): Product containing calories from carbohydrate, protein, and fat
  Interventions: Other: Oral Nutrition Supplement
- Oral Nutrition Supplement D (Active Comparator): Product containing calories from carbohydrate, protein, and fat
  Interventions: Other: Oral Nutrition Supplement
- Oral Nutrition Supplement E (Active Comparator): Product containing calories from carbohydrate, protein, and fat
  Interventions: Other: Oral Nutrition Supplement
- Oral Nutrition Supplement F (Active Comparator): Product containing calories from carbohydrate, protein, and fat
  Interventions: Other: Oral Nutrition Supplement

INTERVENTIONS:
Other: Oral Nutrition Supplement — Product intake of oral nutrition supplement provided

SUMMARY:
This will be a randomized crossover design. The subjects will be randomized to one of six interventions on six separate study days, one week apart.

ELIGIBILITY:
Subject inclusion criteria

All subjects must comply with all the following inclusion criteria:

* Age 20-75 years
* Type 2 diabetes controlled with diet or diet and metformin (Glucophage)
* Hemoglobin A1C less than 9.0%
* Fasting blood glucose less than 180 mg
* Hematocrit levels within normal limits
* Having obtained his/her informed consent

Subject exclusion criteria Subjects representing one or more of the following criteria are excluded from participation in the study.

* Abnormal thyroid function
* Creatinine >2.0 mg/dl
* Potassium <3.5 mEq/l
* Gastrointestinal disease: ulcer, gastritis, diarrhea, gastroparesis, vomiting
* Currently unstable diabetes or under treatment for cancer, heart disease, renal disease
* Unable to give informed consent or follow instructions
* Current insulin therapy or insulin therapy within the past month
* Patient who are pregnant
* Allergies to milk, soy or any component of the test product
* Patient who in the investigators assessment cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial
* Patients with anemia

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose curve (ACU 0-240 minutes) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

SECONDARY OUTCOMES:
Area under the insulin curves (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
Insulinogenic index [Change in Ins30/Change in Glu30] | [Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes]

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No